CLINICAL TRIAL: NCT00005113
Title: An Open-Label, Comparative Study of the Effect of Sirolimus Versus Standard Treatment on Clinical Outcomes and Histologic Progression of Allograft Nephropathy in High Risk Pediatric Renal Transplant Patients
Brief Title: A Study to Compare Treatment With Sirolimus Versus Standard Treatment in Patients Who Have Received a Kidney Transplant
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inability to meet the accrual target of 213.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, William Harmon, Director, Division of Nephrology, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT SRL1; DAIT 0468E1-217-US
Record Dates: First submitted 2000-04-14; First posted 2001-08-31 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: End-Stage Renal Disease; Kidney Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Cyclosporine; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive SRL, CsA/tacrolimus, and corticosteroids for up to 36 months
  Interventions: Drug: Cyclosporine; Drug: Sirolimus; Drug: Tacrolimus
- 2 (Experimental): Participants will receive standard CsA or tacrolimus-based double or triple drug therapy for up to 36 months
  Interventions: Drug: Cyclosporine; Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclosporine — Oral tablet taken daily. Dosage is dependent on weight and is titrated to target trough level.
  Other Names: CsA
Drug: Sirolimus — Dosage in liquid or tablet form is dependent on body surface area and is titrated to target trough level.
  Other Names: SRL
  Arms: 1
Drug: Tacrolimus — dosage is in oral form titrated to target trough level

SUMMARY:
The purpose of this study is to compare treatment with the new drug sirolimus (SRL) versus the standard treatment with cyclosporine (CsA) or tacrolimus in children who have received kidney transplants. SRL is a new medication that may prevent the body's immune system from rejecting organ transplants.

After receiving a kidney transplant, the body recognizes the donated kidney as a foreign invader and triggers the immune system to attack the kidney. This can lead to rejection of the new kidney and a failed transplant. To help reduce the risk of kidney rejection, transplant patients are given immunosuppressant drugs, which reduce the body's normal immune response and allow the transplanted organ to function. CsA or tacrolimus are two drugs that are often given to transplant patients. However, these are powerful drugs, and it can cause serious side effects and put a patient at increased risk for infections. SRL is a new drug that has been shown to reduce a transplant patient's chance of rejecting a new kidney, without serious side effects. This study is necessary to test the safety and effectiveness of SRL in children.

DETAILED DESCRIPTION:
Successful kidney transplantation has gradually improved over the years; much of the improvement has resulted from the use of CsA. However, adequate and tolerable immunosuppression is difficult to achieve with CsA, and rejection episodes are still frequent. CsA is nephrotoxic, with drug toxicity often masking rejection episodes. Other immunosuppressant therapies can result in a range of complications, including metabolic disturbances, adrenocortical insufficiency, and increased risk for infections. Therefore, more effective drugs with less toxicity are needed to prevent acute rejection, especially in the pediatric population where the overall graft survival rate remains significantly lower when compared with that of adult transplant recipients. SRL is an immunosuppressive agent being developed for the prophylaxis of acute renal allograft rejection. SRL has a unique mechanism of action. It inhibits T and B cell activity. In Phase I and II trials in adults, SRL was generally well tolerated and exhibited no apparent nephrotoxic properties, and significantly lower rates of rejection were seen with SRL when compared to placebo.

Patients receive extensive prestudy screening, which includes a renal core biopsy, chest x-ray, bone density study, blood tests, and glomerular filtration rate (GFR). Patients are then randomly assigned to 1 of 2 study treatment groups in a 2:1 ratio (142 patients receive SRL, CsA/tacrolimus, and corticosteroids and 71 patients receive standard CsA or tacrolimus-based double or triple drug therapy). SRL is administered as an oral dose of 3 mg/m2/day. Patients are followed for 3 years on therapy, and then for 1 month of follow-up. A renal core biopsy is performed at the time of study entry and at Months 6, 18, and at early termination of patient in study. Patients undergo physical examinations and various blood tests at specified time intervals during the 37-month study period. Efficacy is assessed by comparing the composite endpoint of biopsy-proven acute rejection, graft loss, or death after 36 months of treatment. Safety is assessed by comparing the composite endpoint of graft loss or death after 36 months of treatment.

ELIGIBILITY:
Inclusion Criteria

Your child may be eligible for this study if he/she:

* Has received a kidney transplant.
* Has experienced 1 or more episodes of acute rejection or chronic rejection; a rejection episode must have responded to treatment and have occurred at least 30 days before study enrollment.
* Has stable kidney function at the time of study enrollment.
* Is 20 years of age or younger.
* Has written informed consent of parent or guardian if under the age of 18.
* Agrees to use birth control during the study and for 3 months following treatment.

Exclusion Criteria

Your child will not be eligible for this study if he/she:

* Has a history of cancer.
* Has received a multi-organ transplant (more than a kidney).
* Has an active infection.
* Has an abnormal chest X-ray.
* Cannot provide a kidney biopsy at time of study entry.
* Is allergic to sirolimus.
* Has received experimental drugs within 4 weeks of study entry.
* Is pregnant.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 1999-07; Primary Completion 2004-07 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of sirolimus | Throughout study

SECONDARY OUTCOMES:
Composite endpoint of biopsy proven acute rejection, graft loss, or death | At Months 6, 12, and 24
Rate of clinically diagnosed acute rejection | At months 6, 12, 24, and 36
Rate of change in glomerular filtration rate | At Month 18
Mean change in volume of allograft fibrosis | At Months 6 and 18
Intragraft expression of cytokines | Throughout study
Cytokine expression and subsequent development of chronic allograft nephropathy | Throughout study

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States